CLINICAL TRIAL: NCT01183936
Title: A Randomised Trial of Surgical Excision Margins for Thick Primary Cutaneous Melanoma (>2 mm). A Multicenter Trial Comparing 2-cm vs 4-cm
Brief Title: Trial of Surgical Excision Margins in Thick Primary Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Cancer Society (Other); Stockholm Cancer Society (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Margins Melanoma; Country specific (Other: Swe; Nat Reg Nr, Dk; 5 dig ser nr (8XXXX), Ea; 5 dig ser nr (7XXXX), Ny; 4 dig ser nr (9XXX))
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 1991-06

CONDITIONS: Melanoma; Surgery; Treatment Outcome
Keywords: Melanoma/mortality/pathology/*surgery; Randomized Controlled Trials as Topic; Survival; Disease-Free Survival
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 cm margin of excision (Active Comparator): Patients with CMM >2 mm treated with an excision of 2-cm.
  Interventions: Procedure: 2-cm margin
- 4 cm margin of excision (Active Comparator): Patients with CMM >2 mm treated with an excision of 4-cm.
  Interventions: Procedure: 4-cm margin

INTERVENTIONS:
Procedure: 2-cm margin — Patients with CMM treated with a surgical safety margin of 2-cm in the surrounding skin and down to the fascia.
  Arms: 2 cm margin of excision
Procedure: 4-cm margin — Patients with CMM treated with a surgical safety margin of 4-cm in the surrounding skin and down to the fascia.
  Arms: 4 cm margin of excision

SUMMARY:
Objectives: The purpose of this study was to assess the effects of an excision margin of 2 cm versus 4 cm for patients with primary cutaneous malignant melanoma (CMM).

Study hypothesis: The hypothesis is that there is no difference between the two treatment arms measured as overall survival and recurrence free survival.

DETAILED DESCRIPTION:
Traditionally CMM have been excised with wide resection margins of 5-cm (sometimes with 10-cm towards the local lymph node basin) with the radical removal of lymph nodes. This treatment emerged from a recommendation from Handley in 1907 based on a single pathological specimen. This "radical" surgical management resulted in bad cosmetic results, lymph oedema, long hospital inpatient stay, frequent skin grafting and/or complicated skin flap reconstructions. Not until some 60-plus years later did questions arise in clinical practices whether the need for this extensive surgery was mandated and clinical practice was not substantially changed until the late 1980's. Retrospective studies published in the 1980s suggested that narrower excision margins may be appropriate for treatment of some CMMs, especially thinner lesions.

Breslow tumour thickness of the CMM is the most important prognostic indicator of localised disease and is therefore the information upon which today's surgical strategies are founded. However, recommendations vary over the world especially for thicker tumors. For CMM of ≤ 1 mm thickness most centers use a 1 cm margin, but for tumours 1.01 - 4 mm the margins of resection are 1-3 cm depending on the country. Most patients with CMM > 4 mm are operated on with a margin of 2-cm today. The different national guidelines are thus, somewhat confusing and in a report from 2004 Thomas showed that a 1-cm margin for CMM with a poor prognosis (≥2 mm) is associated with a greater risk of regional recurrence than in a 3-cm margin, but with a similar survival rate.

Still, quite sound evidence now exists to state that narrower excisions - for thinner tumors - is as safe as more wide surgery. To date, five published randomised trials (11 reports) have been published to access what type of surgery to recommend in the different prognostic groups but despite this effort there are still controversies. In a report by Lens based on 4 randomised trials the authors concluded that current evidence was not sufficient to address the optimal surgical margins for all CMM. Furthermore the Cochrane report from 2009 states; "Current randomised trial evidence is insufficient to address optimal excision margins for primary cutaneous melanoma". However, the studies were not designed to access "optimal" surgery, they were designed to compare one surgical strategy with another, where after the results have been interpreted into clinical guidelines.

In conclusion there is a need for additional studies and further research is required especially for the patients with poorer prognoses, i.e. with tumors >2 mm.

In 1992 a multicenter trial was launched from the Swedish Melanoma Study Group. The 936 patients in the study were included from January 22 1992 to May 19 2004. Patients were recruited from Sweden ( 6 centres with 644 pat), Denmark (180 pat), Estonia (80 pat) and Norway (32 pat). Randomisation routines were set up by the steering committee and eligible patients were randomised locally by telephone calls to national and international cancer centres (upon a histologically proven diagnoses and signed patient consent form). Only patients with a CMM >2 mm and with localised disease (who fulfilled the in- and exclusion criteria) were eligible for study inclusion. Patients with CMM on the hands, feet, head-neck and ano-genital region were excluded. Final surgery must had been planned within 8 weeks after date of diagnosis. All analyses were conducted according to the intention-to-treat principle.

Patients were followed clinically every 3 months for 2 years and thereafter every 6 months up to 5 years. Follow-up data was thus collected from cancer registries, cause of death registries and medical records. The overall mean follow-up time was 6 years and 9 months (6 years and 7 months vs. 6 years and 10 months).

Statistical analyses were made by Kaplan Meier life-table curves. Prognostic factors was assessed with the use of a uni- and multivariate Cox regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Melanoma >2 mm
* Age ≤ 75 yr
* Patients operated on with ≤ 2-cm at diagnosis
* Final surgery planned within 8 weeks after date of diagnosis
* Patient fit for surgery
* Signed patient consent form

Exclusion Criteria:

* Melanoma on hand, foot, head-neck or ano-genital regions
* The presence of in-transit- regional and/or distant spread of the disease
* Illness making patient unfit for surgery
* Previous malignancies except basal cell- and in-situ colli uteri cancer

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 936 (Actual)
Dates: Start 1992-01; Primary Completion 2004-05 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Recurrence free survival

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Ringborg, M.D., Ph.D., Study Director — Dept of Oncology-Pathology, Karolinska Institute

REFERENCES:
- [Derived] Gillgren P, Drzewiecki KT, Niin M, Gullestad HP, Hellborg H, Mansson-Brahme E, Ingvar C, Ringborg U. 2-cm versus 4-cm surgical excision margins for primary cutaneous melanoma thicker than 2 mm: a randomised, multicentre trial. Lancet. 2011 Nov 5;378(9803):1635-42. doi: 10.1016/S0140-6736(11)61546-8. Epub 2011 Oct 23. PMID 22027547